CLINICAL TRIAL: NCT04777669
Title: Removing Background Talker Noise for Cochlear Implant Users
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: York Sound Inc (Industry)
Collaborators: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: SBIR01
Record Dates: First submitted 2021-02-25; First posted 2021-03-02 (Actual); Last update posted 2022-07-12 (Actual); Status verified 2022-07

CONDITIONS: Hearing Loss
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experiment (Experimental): Subjects will be tested for their ability to understand speech with and without noise reduction
  Interventions: Other: Noise Reduction

INTERVENTIONS:
Other: Noise Reduction — In within subject design, listeners will have background noise removed by a noise reduction algorithm

SUMMARY:
When hearing-impaired listeners are properly aided with a hearing aid (HA) or cochlear implant (CI), they are often able to comfortably maintain a conversation in quiet environments. However, in group environments, such as a large family dinner, restaurant, or other environment where multiple people are talking simultaneously, hearing-impaired listeners have great difficulty participating in conversations and frequently withdraw or avoid the situation. As such, it would be highly beneficial to implement an algorithm into HAs or CIs to remove background talkers ("babble") from the signal to reduce listening effort for the hearing-impaired listener and allow them to converse as if they were in a quiet environment. Although HAs and CIs frequently incorporate noise reduction algorithms, these algorithms are not effective when the background is babble. The problem of removing babble involves segregating speech from speech. Hence, the spectral properties of the signal and noise are extremely similar.

Despite these challenges, we developed an algorithm to remove background babble. In the following study will test the ability of cochlear implant users to understand speech with background babble noise using our noise reduction algorithm or no noise reduction algorithm. We hypothesize that CI users will be able to understand significantly more speech in babble noise when using our algorithm.

ELIGIBILITY:
Inclusion Criteria:

Subjects with CIs 12 years of age and older with no diagnosis of other communicative or cognitive disorders. Subjects must have native or native-like English proficiency.

Exclusion Criteria:

No diagnosed cognitive or communicative disorders (other than hearing loss), presence of acute/chronic otitis media, useable acoustic hearing, and non-English speaking.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-04-25 (Actual); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Speech Recognition | 1 day
  The % of words correctly understood in various noisy situations will be measured

CONTACTS AND LOCATIONS:
Locations (1):
- New York University School of Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Data requests will be considered on a case by case basis